CLINICAL TRIAL: NCT02909010
Title: Bispectral Index Monitoring To Guide Sedation In Patients With Non-Neurological Pathology Over 65 Years, Admitted To Intensive Care Unit: Randomized Control Trial
Brief Title: Bispectral Index Monitoring To Guide Sedation In The Critical Care Setting
Acronym: BIS65
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Sofia Contreras Medina, Intensivist, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AC063/15
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Deep Sedation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIS™ Brain Monitoring System (Active Comparator): BIS monitoring to adjust sedation in order to maintain values between 50-60
  Interventions: Device: BIS™ Brain Monitoring System
- RASS Monitorization (Placebo Comparator): sedation was adjusted with the exclusive useof Richmond Agitation-Sedation Scale (RASS) to maintain RASS -2.
  Interventions: Other: RASS

INTERVENTIONS:
Device: BIS™ Brain Monitoring System — The intervention group using BIS monitoring to adjust sedation in order to maintain values between 50-60
  Arms: BIS™ Brain Monitoring System
Other: RASS — control group in which sedation was adjusted with the exclusive use of Richmond Agitation-Sedation Scale (RASS) to maintain RASS -2
  Arms: RASS Monitorization

SUMMARY:
A randomized, control trial to compare the total dose of sedatives use in patients over 65 years admitted to the intensive care unit, guiding sedation by monitoring with BIS® versus monitoring with the exclusive use of sedation scales.

The study will include all patients over 65 years who enter the intensive care unit of the University Hospital of Bellvitge affected with medical or surgical pathology of non neurological etiology who require sedation for more than 24 hours to maintain adaptation to mechanical ventilation.

DETAILED DESCRIPTION:
Patients admitted to the intensive care unit (ICU) usually require use of hypnotics and sedatives to ensure comfort and proper adaptation to mechanical ventilation. An important requirement for an adequate sedation is frequent and proper assessment of its depth. Inadequate sedation can lead to problems of over-sedation, under-sedation and/or delirium in ICU, especially in elderly patients. The main objective od the study is To compare the total dose of sedative use and the rate of over-sedation in patients over 65 years admitted to the ICU, adjusting sedation by monitoring with BIS® versus monitoring with the exclusive use of sedation scales. METHODS. A randomized, clinical trial including patients over 65 years who were admitted to the ICU affected with medical or surgical pathology of non neurological etiology who required sedation for more than 24 hours to maintain adaptation to mechanical ventilation. Patients were randomized into two groups: the intervention group using BIS monitoring to adjust sedation in order to maintain values between 50-60 and; the control group in which sedation was adjusted with the exclusive use of Richmond Agitation-Sedation Scale (RASS) to maintain RASS -2. The study was approved by the institution's Research Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 yers
* Patients admitted to teintensive care unit of the University Hospital of Bellvitge medical or surgical pathology of neurological etiology
* Patiens requiring sedation for more than 24 hours

Exclusion Criteria:

* Patients less than 65 years
* Patients admitted to the ICU with Neurological condition.
* Postoperative patients admitted and extubation is expected within 24 hours.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Total Dose of sedation | Two years
  Total dose of sedatives administered in the intervention group compared with the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Corral, MD, Study Director — Barcelona University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fraser GL, Riker RR. Sedation and analgesia in the critically ill adult. Curr Opin Anaesthesiol. 2007 Apr;20(2):119-23. doi: 10.1097/ACO.0b013e32808255b4. PMID 17413394
- [Background] Carrasco G. Instruments for monitoring intensive care unit sedation. Crit Care. 2000;4(4):217-25. doi: 10.1186/cc697. Epub 2000 Jul 13. PMID 11094504
- [Background] De Deyne C, Struys M, Decruyenaere J, Creupelandt J, Hoste E, Colardyn F. Use of continuous bispectral EEG monitoring to assess depth of sedation in ICU patients. Intensive Care Med. 1998 Dec;24(12):1294-8. doi: 10.1007/s001340050765. PMID 9885883